CLINICAL TRIAL: NCT00798889
Title: A Treatment Protocol For Patients Continuing From A Prior SU011248 Protocol
Brief Title: Rollover Protocol for Prior SU011248 Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181030; NCT00569725 (obsolete NCT alias)
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2012-12

CONDITIONS: Solid Tumors
Keywords: Solid tumors
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib dose varies according to the doses allowed in previous protocol. It is given once a day, orally with various schedules depending on the parent protocol

SUMMARY:
The objective of this protocol is to provide SU011248 treatment for patients who have participated in a SU011248 protocol and are eligible to enter this protocol

ELIGIBILITY:
Inclusion Criteria:

* Prior SU011248 Protocol.
* Eligible to continue SU011248 treatment.

Exclusion Criteria:

* Uncontrolled CNS metastasis.
* Unfit to receive SU011248.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2004-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (29):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albuqurque, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Madison, Wisconsin
- Australia (3):
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, East Melbourne, Victoria
  - Pfizer Investigational Site, Heidelberg, Victoria
- Pfizer Investigational Site, Montreal, Quebec, Canada
- Pfizer Investigational Site, Villejuif, France
- Pfizer Investigational Site, Thessaloniki, Greece
- Pfizer Investigational Site, Milan, Italy
- Pfizer Investigational Site, Nijmegen, Gelderland, Netherlands
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- Sweden (2):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site, Sankt Gallen, Switzerland
- United Kingdom (3):
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Newcastle upon Tyne

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181030&StudyName=Rollover%20Protocol%20for%20Prior%20SU011248%20Protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from prior studies in which they received sunitinib.
Groups:
- Sunitinib: Sunitinib 50 milligram (mg) capsule orally once daily in schedule 4/2 (4 weeks on treatment, 2 weeks off treatment) or schedule 2/1 (2 weeks on treatment, 1 week off treatment) or Schedule 2/2 (2 weeks on treatment, 2 weeks off treatment) or continuous dosing, based on investigator's discretion.
Period: Overall Study
Arm/Group | Sunitinib
Started | 314
Treated | 311
Completed | 0
Not Completed | 314
Not completed — Adverse Event | 53
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 31
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 213
Not completed — Decision of Sponsor | 11
Not completed — Enrolled, Not treated | 3

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib: Sunitinib 50 mg capsule orally once daily in schedule 4/2 (4 weeks on treatment, 2 weeks off treatment) or schedule 2/1 (2 weeks on treatment, 1 week off treatment) or Schedule 2/2 (2 weeks on treatment, 2 weeks off treatment) or continuous dosing, based on investigator's discretion.
Arm/Group | Sunitinib
Number analyzed (Participants) | 311
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 198

OUTCOME MEASURES:

1. Primary Outcome: Duration of Treatment
Time Frame: Baseline up to Day 28 after last dose of study treatment
Population: The intent-to-treat population included all participants who were enrolled in the study and received at least 1 dose of study medication.
Measure: Median (Full Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 311
Days | 190 [3 to 2289]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 118/311
Other Adverse Events (participants affected / at risk) | 299/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=311)
Abdominal pain (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 7
Pancreatitis (Gastrointestinal disorders) | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Caecitis (Gastrointestinal disorders) | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectal obstruction (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 4
Infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Liver abscess (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infectious peritonitis (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Pancreatic abscess (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Disease progression (General disorders) | 9
Pyrexia (General disorders) | 6
Chest pain (General disorders) | 4
Asthenia (General disorders) | 2
Fatigue (General disorders) | 2
Adverse drug reaction (General disorders) | 1
Chest discomfort (General disorders) | 1
Pain (General disorders) | 1
Sudden death (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 13
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Convulsion (Nervous system disorders) | 2
Hepatic encephalopathy (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 4
Hepatic failure (Hepatobiliary disorders) | 4
Cholangitis (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Biliary fistula (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 5
Deep vein thrombosis (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 2
Intra-abdominal haemorrhage (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Arrhythmia (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Arrhythmia supraventricular (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Mental status changes (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=311)
Anaemia (Blood and lymphatic system disorders) | 71
Leukopenia (Blood and lymphatic system disorders) | 32
Neutropenia (Blood and lymphatic system disorders) | 54
Thrombocytopenia (Blood and lymphatic system disorders) | 48
Hypothyroidism (Endocrine disorders) | 39
Periorbital oedema (Eye disorders) | 23
Abdominal discomfort (Gastrointestinal disorders) | 18
Abdominal distension (Gastrointestinal disorders) | 29
Abdominal pain (Gastrointestinal disorders) | 73
Abdominal pain upper (Gastrointestinal disorders) | 41
Constipation (Gastrointestinal disorders) | 66
Diarrhoea (Gastrointestinal disorders) | 179
Dry mouth (Gastrointestinal disorders) | 25
Dyspepsia (Gastrointestinal disorders) | 56
Flatulence (Gastrointestinal disorders) | 31
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 36
Haemorrhoids (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 141
Oral pain (Gastrointestinal disorders) | 34
Stomatitis (Gastrointestinal disorders) | 45
Vomiting (Gastrointestinal disorders) | 93
Asthenia (General disorders) | 23
Chest pain (General disorders) | 29
Chills (General disorders) | 30
Fatigue (General disorders) | 206
Mucosal inflammation (General disorders) | 58
Oedema (General disorders) | 24
Oedema peripheral (General disorders) | 68
Pain (General disorders) | 25
Pyrexia (General disorders) | 60
Sinusitis (Infections and infestations) | 18
Upper respiratory tract infection (Infections and infestations) | 33
Aspartate aminotransferase increased (Investigations) | 16
Blood creatinine increased (Investigations) | 20
Haemoglobin decreased (Investigations) | 20
Weight decreased (Investigations) | 28
Decreased appetite (Metabolism and nutrition disorders) | 103
Dehydration (Metabolism and nutrition disorders) | 25
Hyperglycaemia (Metabolism and nutrition disorders) | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 55
Back pain (Musculoskeletal and connective tissue disorders) | 65
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 64
Dizziness (Nervous system disorders) | 39
Dysgeusia (Nervous system disorders) | 48
Headache (Nervous system disorders) | 73
Neuropathy peripheral (Nervous system disorders) | 25
Peripheral sensory neuropathy (Nervous system disorders) | 16
Anxiety (Psychiatric disorders) | 24
Depression (Psychiatric disorders) | 21
Insomnia (Psychiatric disorders) | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 73
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 79
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 36
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25
Dry skin (Skin and subcutaneous tissue disorders) | 35
Erythema (Skin and subcutaneous tissue disorders) | 19
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 81
Pruritus (Skin and subcutaneous tissue disorders) | 19
Rash (Skin and subcutaneous tissue disorders) | 55
Skin discolouration (Skin and subcutaneous tissue disorders) | 58
Skin discolouration (Skin and subcutaneous tissue disorders) | 18
Flushing (Vascular disorders) | 21
Hypertension (Vascular disorders) | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.